CLINICAL TRIAL: NCT02142452
Title: Cardiovascular Health in Postpartum Women Diagnosed With Excessive Gestational Weight Gain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sandra Anping Tsai, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 28810
Record Dates: First submitted 2014-05-08; First posted 2014-05-20 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Pregnancy; Weight Gain
Keywords: Pregnancy; Obesity/Overweight; postpartum; mobile health; cardiovascular disease
MeSH Terms: conditions — Weight Gain; Obesity; Overweight; Cardiovascular Diseases | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- mobile health intervention (Experimental): Behavioral intervention. Women with excessive weight gain in pregnancy will be recruited in their 3rd trimester. They will begin with a 5 week group session on weight management. After they deliver the baby, they will begin receiving text messages supporting behavior change they learned in their 3rd trimester. They will follow up at 6 weeks postpartum and 4 months postpartum.
  Interventions: Behavioral: behavioral intervention
- Control Group (Placebo Comparator): Women will receive usual prenatal care from their OB. Postpartum, they will receive a monthly newsletter relevant to the new mother on her nutrition and physical activity. They will be followed at 6 weeks postpartum and 4 months postpartum.
  Interventions: Other: Usual Prenatal Care

INTERVENTIONS:
Behavioral: behavioral intervention — Behavioral intervention will include a group class for women in their 3rd trimester followed by a mobile texting program to support behavior change postpartum.
  Arms: mobile health intervention
Other: Usual Prenatal Care
  Arms: Control Group

SUMMARY:
The investigators will test the efficacy of a tailored behavioral lifestyle modification program to support cardiovascular health in postpartum women with excessive gestational weight gain. This program will include a mobile health texting component postpartum to support changes in nutrition and physical activity. The investigators will randomize women into either the control arm (usual care) or the intervention (usual care + mobile health program postpartum). The women will be recruited during their 3rd trimester once they have been identified as gaining too much weight according to the 2009 IOM guidelines during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman diagnosed with excessive gestational weight at 24 weeks gestation or later
* Age 18 years or older
* English-speaking, and willing and able to participate in the proposed intervention.

Exclusion Criteria:

* Inability to provide informed consent and/or an inability to speak, read, or understand English
* Primary residence is outside of the immediate catchment area of 10 miles
* Physical or mental challenges that precludes them from exercising or returning for scheduled study follow ups
* Concurrent enrollment in another behavior modification program

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2014-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
BMI (body mass index) | 4 months postpartum
  A mobile Health intervention tailored for the 30 postpartum mother and grounded in behavioral change theory will be associated with significantly more reduction in BMI than 30 women not enrolled in the intervention.

SECONDARY OUTCOMES:
Cardiovascular health metrics | 4 months postpartum
  (1) Examine changes in cardiovascular health metrics (fasting glucose, fasting insulin, and BP) and markers of inflammation (hs-CRP) verses control group (2) We will evaluate changes in perceived nutrition, physical activity, and weight-loss self-efficacy; self-efficacy has been shown to be a direct predictor of behavior (3) measure the effects of breastfeeding support on the length of time a mother breastfeeds verse the control group.
Change in self efficacy score based on behavioral self-efficacy scale | 4 months postpartum
  We will measure changes in pre- and post-intervention self-efficacy of all women in intervention and control arms.
Cardiovascular health metrics | 4 months postpartum
  We will evaluate changes in perceived nutrition, physical activity, and weight-loss self-efficacy; self-efficacy has been shown to be a direct predictor of behavior
Cardiovascular health metric | 4 months postpartum
  Measure the effects of breastfeeding support on the length of time a mother breastfeeds verse the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra A Tsai, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes